CLINICAL TRIAL: NCT03206983
Title: Efficacy of the Canabrava/s Pupil Expansion Device in Cataract Surgery With Small Pupils: The First 30 Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Casa de Misericórdia de Belo Horizonte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-0928-RG
Record Dates: First submitted 2017-05-18; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Small Pupil; Cataract
Keywords: Small pupil
MeSH Terms: conditions — Miosis; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cana's Ring group (Experimental): The device Cana's Ring was used during cataract surgery on these patients.
  Interventions: Device: Cana's Ring

INTERVENTIONS:
Device: Cana's Ring — The device is used during cataract surgery to help dilate small pupils (under 5mm)

SUMMARY:
To evaluate the intraoperative stability, safety and overall efficacy of the Canabrava Ring (AJL - SPAIN) when used to expand pupils with less diameter than 5 mm and pupils with sphincter synechiae.

DETAILED DESCRIPTION:
In this consecutive case series, 30 eyes of 29 patients underwent cataract surgery using a new disposable small-pupil expansion device, Canabrava's Ring (AJL Ophthalmic, Spain). It is the first iris expansion ring produced with indents that do not align with each other in the superior and inferior regions, resulting in a small vertical length (0.4mm) that minimizes risk of endothelial contact. All eyes had poorly preoperatively dilated pupils of less than 5mm. Fifteen eyes had significant infective or traumatic pathology preoperatively. Vertical and horizontal pupil diameters were evaluated pre-, intra- and 1 month postoperatively, and were used to calculate pupil circumference. Intraoperative and postoperative pupil circumference comprised the primary outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* clinical indication for cataract surgery, age of at least 18 years, pupil diameter less than 5mm after dilation with phenylephrine and tropicamide, and lens with any degree of opacity.

Exclusion Criteria:

* eyes unable to perceive light during visual acuity testing, pupils with a diameter greater than 5mm and clear lenses

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 30 days after surgery
  Safety of the material of the device from break, lesion of eye structures and iritis

SECONDARY OUTCOMES:
Stability of the device during surgery | During surgery
  Evaluate whether the device remains stable and attached to the iris during the entire surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Canabrava, MD, Study Chair — Santa Casa de Misericórdia de Belo Horizonte

IPD SHARING:
Plan to Share IPD: No